CLINICAL TRIAL: NCT06286254
Title: Non-interventional Prospective Study of Safety and Efficacy of the Drug Cycloferone® (NTFF "POLYSAN" Ltd., Russia) in Patients with Acute Respiratory Viral Infection At the Outpatient Stage
Brief Title: Study of Safety and Efficacy of the Drug Cycloferone in Patients with Acute Respiratory Viral Infection
Status: Completed | Type: Observational
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CYCL-NTTF-2023
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-02

CONDITIONS: Acute Respiratory Viral Infection
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The control group: Basic therapy of ARVI1 + Cycloferone®. Cycloferone® is administered according to the instruction for medical use: 600 mg (4 tablets) once daily on day 1, 2, 4, 6 and 8.
  Interventions: Drug: Cycloferone
- The test group: Basic therapy of ARVI1 + Arbidol®. Arbidol® is administered according to the instruction for medical use: 200 mg (4 capsules) 4 times/day for 5 days.

INTERVENTIONS:
Drug: Cycloferone — Cycloferone® is administered according to the instruction for medical use: 600 mg (4 tablets) once daily on day 1, 2, 4, 6 and 8.
  Other Names: paracetamol
  Groups: The control group

SUMMARY:
The study will collect the information on clinical effects and safety of the basic therapy of acute respiratory viral infection (ARVI) + Cycloferone® and basic therapy of ARVI1 + Arbidol® in real-life clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged from 18 to 65 years.
2. According to the routine clinical practice, a patient is scheduled to receive the treatment as per one of the following regimens:

   - Basic therapy of ARVI1 + Cycloferone®.
   * Basic therapy of ARVI1 + Arbidol®.
3. Presence of symptoms of ARVI:

   * Presence of two and more symptoms of moderate severity or three and more mild symptoms in accordance with the WURSS-21 questionnaire;
   * Presence of two and more symptoms of moderate severity or three and more mild symptoms in accordance with the CCQ questionnaire;
   * Presence of hyperthermia episodes ≥ 37.5°С and ≤ 40.0°С from onset of the disease.

<!-- -->

1. Male and female patients aged from 18 to 65 years.
2. According to the routine clinical practice, a patient is scheduled to receive the treatment as per one of the following regimens:

   - Basic therapy of ARVI1 + Cycloferone®.

   - Basic therapy of ARVI1 + Arbidol®.
3. Presence of symptoms of ARVI:

   - Presence of two and more symptoms of moderate severity or three and more mild symptoms in accordance with the WURSS-21 questionnaire;
   * Presence of two and more symptoms of moderate severity or three and more mild symptoms in accordance with the CCQ questionnaire;
   * Presence of hyperthermia episodes ≥ 37.5°С and ≤ 40.0°С from onset of the disease.
4. Diagnosis as per ICD-10 (primary diagnosis is one of the below diagnoses):

   - J00 - Acute nasopharyngitis, rhinitis;

   - J02 - Acute pharyngitis;

   - J02.8 - Acute pharyngitis caused by other specified pathogens;

   - J02.9 - Acute pharyngitis, not otherwise specified;

   - J03 - Acute tonsillitis;

   - J03.8 - Acute tonsillitis caused by other specified pathogens;

   - J02.9 - Acute tonsillitis, not otherwise specified;

   - J04 - Acute laryngitis and tracheitis;

   - J04.0 - Acute laryngitis;

   - J04.1 - Acute tracheitis;

   - J04.2 - Acute laryngotracheitis;

   - J05 - Acute obstructive laryngitis (croup);

   - J05.0 - Acute obstructive laryngitis (croup);

   - J06 - Acute infection of the upper respiratory tract of multiple and unspecified localization;

   - J06.0 - Acute laryngopharyngitis;

   - J06.8 - Other acute infections of the upper respiratory tract of multiple localization;

   - J06.9 - Acute infection of the upper respiratory tract, not otherwise specified;

   - J20.4 - Acute bronchitis caused by parainfluenza virus;

   - J20.5 - Acute bronchitis caused respiratory syncitial virus;

   - J20.6 - Acute bronchitis caused by rhinovirus;

   - J20.8 - Acute bronchitis caused by other specified agents;

   - J20.9 - Acute bronchitis, not otherwise specified;

   - J21 - Acute bronchiolitis;

   - J21.0 - Acute bronchiolitis caused by respiratory syncytial virus;

   - J21.8 - Acute bronchiolitis caused by other specified agents;

   - J21.9 - Acute bronchiolitis, not otherwise specified;

   - J22 - Acute respiratory infection of lower respiratory tract, not otherwise specified;

   - B34.0 - Adenovirus infection, not otherwise specified;

   - B34.9 - Viral infection, not otherwise specified;

   - B97.0 - Adenovirus infection;
   * B97.4 - Respiratory syncytial infection.
5. Symptoms of the disease are present for not more than 24 h before inclusion in the study.
6. Patient's written consent for participation in the study.

Exclusion Criteria:

1. The use of other drugs having antiviral and/or immune stimulating and/or immune modulating effect.
2. Positive result of SARS-CoV-2 RNA PCR test.
3. Suspected novel coronavirus infection COVID-19 in accordance with the Temporary Methodical Recommendations of the MoH of RF on Prophylaxis, Diagnostics and Treatment of Novel Coronavirus Infection (COVID-19) (current version at the time of inclusion of patients).
4. Current bacterial infection requiring administration of antibacterial drugs.
5. Active non-respiratory viral infection: meningitis, encephalitis, pneumonitis.
6. Availability of indications for hospitalization.
7. Chronic pulmonary diseases (asthma, chronic obstructive pulmonary disease, cystic fibrosis, pulmonary emphysema, tracheobronchial dyskinesia, bronchiectasis etc.).
8. Pulmonary tuberculosis (active or inactive form).
9. Chronic heart failure of functional classes III-IV according to functional classification of the New York Heart Association (NYHA) including instable progressive angina pectoris of functional class IV, uncontrolled arterial hypertension, severe arterial hypotension, severe arrhythmia requiring the treatment with antiarrhythmic drugs of classes Ia, Ib, Ic or III, myocardial infarction, surgeries on the heart and coronary vessels, transient ischemic attack or stroke, pulmonary embolism or deep vein thrombosis.
10. Psychic diseases, neuromuscular, neurocognitive disorders, history of epilepsy.
11. Decompensated diabetes mellitus.
12. Obesity of degree 2-3 (body mass index ≥ 35.0 kg/m2).
13. Severe decompensated renal and hepatic diseases including cirrhosis (acute/chronic renal/hepatic failure).
14. Thyroid diseases.
15. Stomach and duodenum ulcer or other erosive-ulcerative gastrointestinal disorders in exacerbation stage.
16. Malabsorption syndrome or other clinically significant gastrointestinal disease (uncorrected vomiting, diarrhea, ulcerative colitis and others).
17. Malignant neoplasms.
18. Pregnancy, breast feeding.
19. Hemoglobinopathy.
20. Primary and secondary immunodeficiencies (HIV-infection, use of immunosuppressants, systemic glucocorticoids etc.).
21. Contraindications mentioned in the approved instructions for use of the drugs used in the study.
22. Disease or use of medicines, which, in the doctor's opinion, can influence safety, tolerability and efficiency of the study medicines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptoms of ARVI receiving the therapy at the outpatient stage.
Sampling Method: Probability Sample
Enrollment: 742 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Average fever duration according to the data of the Patient's Diary | Baseline, up to 9 days
  ending of fever is defined as body temperature < 37.0°С for 24 hours and more

SECONDARY OUTCOMES:
Dynamics of symptom severity parameter according to WURSS-21* questionnaire by visit 2, 3 and 4 (AUC value of change in symptom severity according to WURSS-21 questionnaire)** | Baseline, 3 day, 5 day, 9 day
  *Wisconsin Upper Respiratory Symptom Survey - 21. The WURSS-21 is a valid and reliable self-report research tool incorporating specific symptoms and functional impairments common to Acute upper respiratory infection
  **Dynamics of symptom severity according to WURSS-21 scale is assessed using the area under the curve (AUC) at visits 2, 3 and 4. AUC is calculated using the trapezoidal rule. WURSS-21 consists of 21 items (2 questions and 2 domains). Domain of symptoms consists of 10 items: rhinitis, nasal stuffiness, sneezing, sore throat, throat irritation, cough, hoarseness, headache, chest congestion, feeling of fatigue. Domain of abilities consists of 9 items: ability to think clearly, sleep well, breath freely, walk, go upstairs, do physical exercises, fulfil everyday life actions, work not at home, work at home, interact with people, live own private life. The first 20 items are assessed by the 8-point scale (from 0 to 7). The last item is assessed by the 7-point scale (from 0 to
Dynamics of symptom severity parameter according to CCQ scale by visit 2, 3 and 4 | Baseline, 3 day, 5 day, 9 day
  CCQ (Common Cold Questionnaire)
Time (days) till disappearance of disease symptoms according to WURSS-21 scale. | Baseline, 3 day, 5 day, 9 day
  Wisconsin Upper Respiratory Symptom Survey - 21
Number of patients with symptoms of disease and everyday activity disturbance of different severity degree according to WURSS-21 scale. | Baseline, 3 day, 5 day, 9 day
  Wisconsin Upper Respiratory Symptom Survey - 21
Number of patients with symptoms of disease of different severity degree according to CCQ scale. | Baseline, 3 day, 5 day, 9 day
  CCQ (Common Cold Questionnaire)
Number of patients with complete disappearance of symptoms according to WURSS-21 questionnaire per each day of the therapy. | Baseline, 3 day, 5 day, 9 day
  Wisconsin Upper Respiratory Symptom Survey - 21
Frequency of the need to administer the systemic antibacterial therapy | Baseline, 3 day, 5 day, 9 day
  Frequency of the need to administer the systemic antibacterial therapy
Percentage of patients who needed hospitalization | Baseline, 3 day, 5 day, 9 day
  Hospitalization
Average duration of the temporary incapacity period. | Baseline, 3 day, 5 day, 9 day
  Duration of the temporary incapacity period
Frequency of revealing ARVI pathogen before beginning of the therapy (at visit 1) for each pathogen among those patients who underwent the qualitative investigation for ARVI pathogen. | Baseline, 3 day, 5 day, 9 day
  Acute respiratory viral infection (ARVI)
Percentage of patients with negative result of the qualitative investigation for ARVI pathogen by visits 3 and 4 among those patients in whom the pathogen was revealed at visit 1. | Baseline, 3 day, 5 day, 9 day
  Acute respiratory viral infection (ARVI)

CONTACTS AND LOCATIONS:
Locations (13):
- Russia (13):
  - Clinic Zvezdnaya, Saint Petersburg
  - Medical center Astarta, Saint Petersburg
  - Medical Center Energiya Zdoroviy, Saint Petersburg
  - Medical Center Meily, Saint Petersburg
  - Medical Center Oris, Saint Petersburg
  - Medical Center PiterClinica, Saint Petersburg
  - Medical Center Reavita Med, Saint Petersburg
  - Medical Center SOGAZ, Saint Petersburg
  - Research Center Eco-Safety, Saint Petersburg
  - Сity clinic No. 117, Saint Petersburg
  - Сity clinic No. 44, Saint Petersburg
  - Сity clinic No.109, Saint Petersburg
  - Сity hospital No. 40, Sestroretsk

IPD SHARING:
Plan to Share IPD: No